CLINICAL TRIAL: NCT02403934
Title: The Use of Jaw Elevation Device in Deep Sedation
Brief Title: Jaw Elevation Device in Deep Sedation Study
Status: Completed | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NMCSD.2012.0033
Record Dates: First submitted 2015-02-19; First posted 2015-03-31 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Airway Obstruction
Keywords: Airway Management; deep sedation; Jaw elevation device
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Jaw Elevation Device (JED) — apply JED when End tidal O2 low

SUMMARY:
Maintaining a patent airway is a constant concern to any anesthesia provider performing deep sedation cases. The doses of sedative medications often required for the desired level of sedation in a patient often result in occlusion of the airway and the patient becoming apneic. Opening the collapsed or occluded airway requires the use of an invasive airway device, (e.g. laryngeal mask airway (LMA), oral airway or nasal airway) or the application of a jaw thrust maneuver. When the provider provides jaw thrust while attending to the other duties, the patient may not have adequate ventilation and the patient's oxygen saturation can fall producing hypoxemia. Airway management devices currently available require deeper levels of sedation to be tolerated by patients. In order to avoid the need for internal airway devices, providers attempt to carefully adjust the level of sedation so that no airway support is required. For safety, providers usually try to stay on the "light" side of the sedation scale. Unfortunately, this often results in an uncomfortable patient or one who is moving too much to successfully carry out the procedure. Until the availability of the Jaw Elevation Device (JED) there was no external device providers could utilize to assist in opening a patient's airway. By duplicating the jaw thrust maneuver, the JED maintains a patent airway. Once applied, it frees the anesthesia provider to attend to other duties associated with administration of anesthesia without requiring the provider to manually maintain a jaw thrust maneuver. The advantages with such a device would allow a level of sedation deep enough for the patient to tolerate the procedure as well as maintain a patent airway. To date, there have not been any studies evaluating the JED in clinical practice. The investigators wish to evaluate the JED in a standardized fashion during deep sedation or monitored anesthesia care (MAC). Our study would involve 50 patients who became apneic during deep sedation or MAC. A jaw thrust maneuver will be initially performed to demonstrate that each patient's airway can be adequately supported by this maneuver. The JED will then be placed in order to maintain a patent airway, while leaving the level of sedation unchanged. Intraoperative monitoring, continuous ECG, pulse oximetry, blood pressure, capnography, will be routine, and determined by the anesthesia team. The investigators will also track how often the provider was required to adjust the JED to maintain a patent airway, and if the need to convert to an alternate method of airway management was required. The investigators will pursue publication of the results as the first study demonstrating the efficacy of the JED.

DETAILED DESCRIPTION:
1. General Approach: 50 Research subjects will be selected from patients scheduled to undergo transvaginal oocyte (egg) retrieval under sedation or MAC. Sedation for these procedures typically consists of intravenous administration of a combination of midazolam, fentanyl, propofol, and/or ketamine titrated until the patient is calm, while supplemental oxygen is provided by mask or nasal cannula. A continuous infusion of propofol is then begun to keep the patient sedated enough that they will lie still and breathe regularly, but still respond to commands or noxious stimuli (such as a sternal rub). As per standard anesthetic care, each patient will have their oxygen saturation, end-tidal carbon dioxide waveform and heart rate/rhythm measured continuously while the anesthesia care provider monitors the patient for signs of inadequate respiration and airway obstruction. These signs include a loss of the end-tidal carbon dioxide waveform, snoring, paradoxical ventilation, cessation of ventilatory efforts, or a reduction in the oxygen saturation. Typically, whenever these signs are present, the anesthesia provider provides a jaw thrust to open the patient's airway and restore adequate ventilation. Once accomplished, the anesthesia care provider typically lowers the dose of anesthetic and releases jaw thrust. If signs of airway obstruction recur, jaw thrust is applied again until the level of sedation has reached a level low enough that the patient can breathe without airway support. However, this may lead to inadequate sedation, patient movement and difficulty for the surgeon to perform the procedure. The depth of sedation required for the egg retrieval procedure frequently results in needing to perform a jaw thrust or placing an airway device to maintain airway patency. Applying the JED after a jaw thrust may alleviate the airway obstruction while allowing adequate sedation to be maintained without a compromise in the anesthetic depth.

2. Description: Prior to anesthesia, all subjects will be given supplemental oxygen and monitored with pulse oximetry, end tidal carbon dioxide (ETCO2) capnography, noninvasive blood pressure, heart rate and rhythm measurement. In this study, once the patient is sedated and inadequate ventilation is identified as stated above, a jaw thrust maneuver will be applied. If this maintains adequate ventilation the JED will then be placed on the patient and adjusted to produce a simulated jaw thrust in an effort to open the obstructive airway. Once the JED is appropriately placed and clinical signs of ventilation achieved, the investigator will document the number of times that the anesthesia provider must manipulate the JED device to achieve an adequate airway. If at any time the anesthesia care provider feels that the JED cannot be adjusted to successfully maintain the airway, the use of the JED will be discontinued and the anesthesia provider will employ an airway management technique of their choice. In addition, the time of initial placement of the JED until end of JED use will be recorded to obtain total time of JED use during the anesthetic. The number of adjustments per unit time of JED use will then be calculated to compare to a constant jaw thrust that would otherwise be required. The duration of anesthesia administration with also be collected beginning with induction of anesthesia/sedation until cessation of infusion. The study will be continued until 50 patients have been entered into the study. Information will be collected even if the patient does not require a jaw thrust and the JED is not placed. Due to the high frequency of requiring airway assistance with egg retrieval procedures performed under deep sedation, the incidence of patients not requiring assistance is likely to be low and 50 patients was felt to be an adequate study size to describe the utility and efficacy of the JED in this setting.

3 Methods: One of the above listed investigators will observe the anesthetic and collect observed data listed on the attached data collection sheet. Data to be collected will include the following:

Data point Method of measurement Date of procedure day/month/year (DD/MM/YYYY) Patient gender Population is all female ASA class 1-6 Age In years Height inches Weight kilograms BMI Kg/m2 Patient ethnicity How patient identifies Patient history of obstructive sleep apne (OSA) Asked pre-operatively STOP-BANG score Asked pre-operatively Patient diagnosis Infertility Duration of anesthetic medication administration Minutes:seconds Medication used Name of medication Medication dose Mg, mcg Medication infusion rate Mcg/kg/min Time from initiation of sedation to first airway obstruction Minutes:seconds Obstruction relieved with jaw thrust Yes/No Success of JED placement Return of patent airway Time from JED placement to next airway manipulation, Minutes:seconds Number of airway manipulations required after JED placement counting Frequency of hypoxemia arterial oxygen saturation (SaO2) <90% Duration of hypoxemia Minutes:seconds Complications List complications Conversion to GA Yes/No Method of GA List method Other airway devices used List device

4. Investigational Drugs/Devices/Biologics Research: Jaw Elevation Device (JED). The FDA has determined the JED is a Class 1 device and thus exempt from 510 K.

5. Research Material Collected: A data collection form will be filled out by the anesthesia provider and returned to an investigator. Information will include details about the anesthetic technique used, and the performance of the JED.

6. Protection of Patient Privacy: All documents relating to an individual's participation in this study will be kept in a locked storage. Access to records will be limited to the PI and AI's. Computer files containing collected study data will be stored in a password protected file system. Identifying information will be recorded on separate form and linked to data collection forms with a numbering system, deidentifying the data. Data will be transcribed into secured electronic files which will be used for data analysis. Once data analysis is complete the data collection sheets will be destroyed or shredded.

7. Risks: This study confers no additional risk to patients as this in an observational study using the JED in a marketed application. All patients in the study will receive the same treatment. There are associated risks with receiving deep sedation. These include but are not limited to: airway obstruction, need to use other types of airway devices including an endotracheal tube, sore throat, nausea and vomiting, aspiration, and other serious, but rare, complications (cardiovascular or pulmonary complications). However, these are risks inherent to the administration of sedation for your procedure. You would be at risk for these whether or not you participated in this study.

8. Radiation or Laser Exposure: None

9. Justification of Risks: The JED offers the potential advantage of increasing the range of patients who could safely tolerate deep sedation or MAC. By completing this study we hope to begin the characterization of populations who can benefit from the use of JED in deep sedation or MAC.

10. Minimization of Risks: By providing a systematic approach to patient selection and data collection we hope to gain maximum utility from our study. By performing this study in an observational fashion we will allow anesthesia providers to retain full control of anesthetic management, for essentially no alteration in the standard of care, and virtually no additional clinical risk. Risk of the exposure of PHI will minimized through the methods discussed above.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients undergoing egg retrieval for infertility requiring deep sedation or MAC and
* who can lie in the supine position throughout the entire procedure.

Exclusion Criteria:

* Adult female patients who are known to have allergies or intolerances to the intended sedative medications that will be used as the primary anesthetic and
* patients who have an upper airway, facial, or jaw anatomic abnormality that the anesthesia provider determines would be inappropriate to use the JED.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult female patients undergoing egg retrieval for infertility requiring deep sedation or MAC as their anesthetic method.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of a new external airway support device, the JED, when used during deep sedation or MAC in women undergoing egg retrieval. # of air way obstructions (Measured Sa02<90%) | Number of Minutes from start of procedure to end of procedure up to 100 minutes

SECONDARY OUTCOMES:
Change from deep anesthesia to general anesthesia | Number of minutes from start of procedure to end of procedure up to 100 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Judd Whiting, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- NMCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No